CLINICAL TRIAL: NCT04217642
Title: Hip Fracture Cohort in Cauca: Factors That Delay Surgery and Its Outcomes.
Brief Title: Hip Fracture in Cauca. Cohort Study
Acronym: HIPCCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad del Cauca (Other)
Collaborators: Hospital Universitario San José (Unknown)
Responsible Party: Principal Investigator, Angela Maria Merchan, Principal investigator, Universidad del Cauca
Other Study IDs: 5231
Record Dates: First submitted 2020-01-01; First posted 2020-01-03 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hip Fractures
Keywords: Hip fractures; Delay surgery; Quality of life; Outcomes
MeSH Terms: conditions — Hip Fractures | interventions — Fracture Fixation, Internal; Hemiarthroplasty; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delay surgery: Patients who have passed more than 48 hours from admission to surgery
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — The specific surgical technique -osteosynthesis, hemiarthroplasty, or total hip arthroplasty- will depend on the characteristics of the proximal femur fracture in each patient.
  Other Names: Hemiarthroplasty; Total hip arthroplasty

SUMMARY:
This research project is an observational, analytical, prospective cohort study, which aims to identify and describe the causes of delay in surgical intervention in patients with a diagnosis of hip fracture at Hospital Universitario San José, correlate those factors with complications , the impact of the quality of life and the main outcomes in relation to morbidity and mortality associated with the delay in surgery in the study population.

In order to carry out this investigation, the recruitment of patients over 18 years old, who enter our institution with a diagnosis of hip fracture, prior acceptance by the patient or his family member to participate through an informed consent signature is carried out. Subsequently, the research team consults the medical history to monitor the factors that influence the time from admission to surgery. A survey is also conducted to assess the quality of life and how your health status can affect it; which is performed during the hospital stay before surgery, the third day after surgery, one month and 6 months later, the last two surveys are conducted in the control consultation with the treatment team or by call telephone.

It is clear that this study does not represent any risk for the participants, the information collected will be confidential and will not be used for any other purpose outside the investigation.

DETAILED DESCRIPTION:
Hip fracture is an important cause of disability, functional risk and death in the adult population, being more significant in the elderly, it also entails high costs for the health system. Although it is usually rare before the sixth decade of life and is very rare in young people, patients who present a hip fracture functional risk can be very important, reaching prostration in up to 8% of cases when Your surgical management is delayed. It is known that the time elapsed between diagnosis and treatment that affects the survival of patients, because every two days of surgical waiting doubles the probability of death due to secondary complications such as infections and cardiovascular complications, which impacts on flexibility and quality. of the patient's life. In addition, it should be borne in mind that in occasions it is necessary to stabilize chronic pathologies of the patient, preventing this sea intervened in a timely manner.

At present there is no consensus on the intervention time of these fractures; However, previous studies have found that better results are obtained when surgical treatment is performed within the first 24 hours. In Colombia there are few published studies describing epidemiological characteristics, estimated time from admission to the surgical procedure, and the factors that specific to such delay. Due to the above and considering that hip fracture is considered a public health problem, it is important to identify sociodemographic factors and medical conditions that may be related to the postoperative complications, morbidity and mortality of these patients to help with the taking of therapeutic and administrative decisions that lead to improving the care provided and final results in the patient.

The general objective of this study is to identify the main causes of delay in surgical intervention in patients with a diagnosis of hip fracture of the San José university hospital during 2019 and its relationship with morbidity and mortality.

The research team has also proposed the following specific objectives to carry out this study:

1. Describe socio-demographically the patients with a diagnosis of hip fracture, underwent surgery at the San José University hospital since 2019.
2. Identify the reason that delay in surgical intervention.
3. Quantify the main outcomes in morbidity and mortality during the 6 months after surgery, associated with the delay in surgery in the study population.
4. Assess the quality of post-surgical life in the patient operated on for hip fracture.
5. Correlate the delay in surgical intervention with complications and mortality in patients operated for hip fracture since 2019.

It is estimated to include 80 patients during the first year of recruitment. For the collection of information there is a sociodemographic survey, the EQ5D5L quality of life survey and comorbidity is evaluated taking into account the Charlson index.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or female) ≥ 18 years of age
* Diagnosis of femoral fracture
* Receiving surgical treatment

Exclusion Criteria:

* Patients with cognitive disorders that prevent interrogation and assessment of quality of life.
* Patients referred to another institution for surgery.
* Patient who decides to voluntarily withdraw from the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized at the San José de Popayán University Hospital for surgical correction of hip fractures that meet the inclusion criteria since 2019. Written informed consent will be obtained from all patients.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Delay surgery | 1 month
  Time, in hours, from emergency room admission until surgery.

SECONDARY OUTCOMES:
QoL | 12 months
  Quality of life whit the 5-level EQ-5D version (EQ-5D-5L generic questionnaire by EuroQol) assessed preoperatively and postoperatively at days 5 and 30 and months 6 and 12.
  The EQ-5D-5L measures 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) related to quality of life. Each dimension has 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and extreme problems) which are scored from 1 (no problems) to 5 (extreme problems) points, with the maximum score of 1 indicating a state of full health.
Mortality | 12 months
  All causes mortality

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Merchán Galvis, MD, MSc, Principal Investigator — Universidad del Cauca
Locations (1):
- Hospital Universitario San José, Popayán, Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Merchan-Galvis AM, Munoz-Garcia DA, Solano F, Velasquez JC, Sotelo NF, Molina DA, Caicedo JP, Concha JM, Calvache JA, Martinez-Zapata MJ. Delayed surgery and health related quality of life in patients with proximal femoral fracture. Sci Rep. 2023 Jul 10;13(1):11131. doi: 10.1038/s41598-023-33592-3. PMID 37429947